CLINICAL TRIAL: NCT05523076
Title: Transdiagnostic Markers of Cognitive Symptoms in Disorders Affective.
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other); Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Maria J Portella, Head of the Research Group in Psychiatric Disorders, Hospital de Sant Pau, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-AFE-2018-10
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; BDMF; GSH; Neurologic Manifestations
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sampling of peripheral inflammatory markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this project is to determine the concordance between the subjective and objective evaluation of cognitive functions in affective patients in partial remission through scales and cognitive tests that would be easily implemented in the different mental health care devices.

This is a cross-sectional case-control study of non-probabilistic sampling, which will include a group of patients diagnosed with Major Depressive Disorder and Bipolar Disorder and a group of healthy controls from the same population and matched by age, gender and years of education with the group of patients.

Patients will be recruited from the psychiatric service of the Hospital de la Santa Creu i Sant Pau who meet the inclusion criteria, and they will undergo a blood draw, a clinical assessment, a complete neuropsychological examination together with scales of subjective perception of cognitive deficit, a measure of cognitive reserve and an evaluation of psychosocial functionality. In addition, the same evaluation will be made to a group of healthy subjects.The total sample will be 120

DETAILED DESCRIPTION:
This is a cross-sectional study with the following hypotheses and objectives:

1. Patients will show an objective cognitive deficit with both subjective and objective measures compared to healthy controls.
2. Subjectively and objectively assessed cognitive deficits will show moderate agreement in patients with a depressive episode in partial remission, as each assesses different aspects of cognition.
3. Both the subjective and the objective assessment will have a high agreement between patients with DM and TB, demonstrating the transdiagnostic nature of self-assessed and heteroassessed cognitive deficits.
4. Cognitive Reserve will be a mediating factor in the correlation between subjective and objective cognitive evaluation.
5. BDNF and GSH will be associated with the patients' cognitive deficit and will act as mediators between the subjective and objective assessment.

Main Objective:

To study the impact of cognitive reserve and trophic factors and oxidative stress as transdiagnostic markers of cognitive symptoms (subjective and objective) in patients with DM and TB.

1. Cognitively assess patients with DM and TB (in a depressive episode) through subjective assessment and objective assessment.
2. Evaluate the possible implementation of objective (SCIP) and subjective (COBRA, PDQ) cognitive assessment instruments.
3. Determine the degree of agreement between both types of cognitive assessment both intra-patient and inter-diagnostic.
4. Determine the factors associated with the degree of agreement between both assessments (Cognitive Reserve, BDNF and GSH) in and between both affective disorders.

ELIGIBILITY:
Inclusion Criteria:

* 8 and 60 years (males and females)
* diagnosis of Major Depression (criteria Diagnostic and Statistical Manual 5th edition, DSM-5) in Remission or Partial Remission phase (scores below 14 in the Hamilton Depression Rating Scale-17 items (HDRS-17))
* Cognitive Symptoms (-1.5SD (standar deviation) in objective as subjective tests)
* PDQ > 20
* FAST> 17

Exclusion Criteria:

* Intelligence Quotient (IQ) < 85
* Any medical condition that may affect cognition
* Presence of any comorbid psychiatric condition (including abuse or dependence on substances in the last three months)
* Electroconvulsive therapy (ECT) in the previous year
* Other psychological intervention in the 6 months prior to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be patients with major depressive disorder and bipolar disorder. In addition, a control group with healthy subjects matched by age, educational level and sex will be included.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive outcome | 1 assessment
  Composite score of different neuropsychological tests

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain